CLINICAL TRIAL: NCT06290297
Title: Assessment and Telerehabilitation of Cognitive and Motor Skills in Children With Neurodevelopmental Disabilities
Brief Title: Assessment and Telerehabilitation of Cognitive and Motor Skills in Children With Neurodevelopmental Disabilities (Tablet Project)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus (Other); IRCCS Eugenio Medea (Other); Oasi Research Institute-IRCCS (Other); Ospedale Pediatrico Bambin Gesù (Other); IRCCS San Raffaele Roma (Other); IRCCS National Neurological Institute "C. Mondino" Foundation (Other); IRCCS Centro Neurolesi Bonino Pulejo (Other); Istituto Giannina Gaslini (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); IRCCS Ospedale San Raffaele (Other); IRCCS Istituto delle Scienze Neurologiche di Bologna (Other)
Responsible Party: Principal Investigator, Giuseppina Sgandurra, MD, PhD, IRCCS Fondazione Stella Maris
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Progetti di Rete (RIN-IDEA)
Record Dates: First submitted 2024-02-16; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Neurodevelopmental Cognitive, Motor and Speech-language Disabilities
Keywords: Neurodevelopmental disabilities; cognitive functions; motor skills; telerehabilitation; technologies; speech functions; ICTs; innovation; congenital and acquired disabilities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with neurodevelopmental disabilities (Experimental): Children aged 4 to 18 with cognitive, motor and/or speech-language impairments
  Interventions: Device: Telerehabilitation VRRS

INTERVENTIONS:
Device: Telerehabilitation VRRS — Telerehabilitation programs delivered at home, aiming to improve cognitive, motor and/or speech-language skills, through VRRS - Khymeia or Niurion devices. Such technologies are equipped with a wide library of activities to be performed also with the use of peripheral sensors. A one-shot assessment is also proposed to children admitted to institutes adhering to the project in order to understand the feasibility of the use of such devices. Ad hoc feasibility questionnaire are administered at the end of the one shot session and after the home training to the main stakeholders (children, families, clinicians)

SUMMARY:
The development and application of new technologies to support functional assessment and rehabilitation pathways for neurodevelopmental disabilities allow the evaluation and enhancement of cognitive, motor, and speech abilities within a more playful and motivating context. In fact telerehabilitation programs foster access to rehabilitative services and permit the delivery of a wide range of neuropsychological, motor, speech and communication interventions, even for patients unable to frequently attend a clinical institution (distance from the hospital, parental work employment, etc.), by overcoming geographic barriers. In this scenario, new technologies guarantee significant time- and cost-saving, shortening hospitalization and delivering the rehabilitative process at home, in a more ecological context (American Telemedicine Association, 2017) therefore enforcing the generalization of the achieved competences. Another great advantage provided by using innovative technologies in clinical practice to foster therapies tailored to patient's needs concerns both the possibility of collecting comprehensive and accurate quantitative data, thus supporting a better intervention monitoring, and of offering multi domain activities, also integrating peripheral devices (i.e. sensors). Using innovative technologies in clinical practice also give the possibility to propose neuropsychological and motor activities in a playful and motivating context, thus enhancing participation and enjoyment, especially for the pediatric population, while maintaining high levels of efficiency. Such telerehabilitation pathways allow to increase dosage and intensity of the intervention and ensure caregivers' involvement in the rehabilitation process. This multicenter study aims to assess the feasibility of using technological systems, primarily validated in the adult population, in children with congenital and acquired disabilities by administering ad-hoc questionnaires.

DETAILED DESCRIPTION:
The study aims assessing the feasibility of using technological systems, in a pediatric population with congenital and acquired neurodevelopmental disabilities, for the assessment and rehabilitation of cognitive, motor and speech functions. A group of children aged between 4 and 18 years with neurodevelopmental disabilities of heterogeneous etiopathogenesis is selected. A non-randomized allocation is planned based on the specific children needs, according to their age and functional profile.

Specifically, the study has envisaged several detailed phases. At first, an analysis of the exercises within the library of the technological systems used by participating IRCCS (VRRS - Khymeia, Niurion) is conducted. After a careful evaluation, the selected exercises (based on age and functional profile) are categorized using a rating methodology and expert discussions, in order to identify specific protocols according to the involved cognitive, speech, and/or motor function. Options for the different exercises are discussed and organized to order them hierarchically and plan a progression of activity proposals based on required skill levels. Some implementation of the present exercises are proposed, in order to make the system more suitable for developmental age, thanks to the collaboration between the clinical staff and the producers.

The created protocols are administered as one-shot assessment in a single session to a group of 4-18 years old children with neurodevelopmental disabilities. Usability and acceptability questionnaires, specifically created for this purpose, are administered, to assess the feasibility of using such technological systems, validated for adults, in the pediatric population. According to the functional profile and one-shot session the possibility of undergoing a tele-rehabilitation program is also considered for each child, with variable duration and frequency based on specific children and caregivers emerging needs. Specific inclusion and exclusion criteria are defined:

Inclusion Age between 4-18 years old Non-degenerative, congenital or acquired neurodevelopmental disability A cognitive functioning sufficient for understanding instructions and participating in delivered activities MACS <5 Exclusion Severe associated pathologies Criteria for the accessibility to tele-rehabilitation programs are also established, including a distance from the clinical center to allow periodic in-person evaluation of the training progress, internet access availability, and the willingness of parents and/or legal guardians to engage in and collaborate with an intensive home-based rehabilitation program.

Participants included in a tele-rehabilitation intervention (cognitive, motor, speech, or integrated) are provided with ICT technologies, delivered directly to their homes, including peripheral devices and a user manual for caregivers. Rehabilitation sessions at home are constantly monitored remotely by the rehabilitation staff, either online or through the offline viewing of obtained reports. Intervention has a global duration of 30 sessions at least, with a variable frequency based on specific children and caregivers emerging needs.

Finally, indicators for measuring the feasibility and effectiveness of different tele-rehabilitation programs are selected based on the literature, as well as clinical assessment scales for cognitive, speech and motor skills. Questionnaires for each end-user category have been developed to analyze different aspects of usability and acceptability, including perceived satisfaction, effectiveness, and efficiency on one hand, and experienced ease of use and utility on the other. From a clinical perspective, a shared protocol of pre-post training clinical measures has been developed to evaluate not only specific cognitive, speech and motor aspects but also any impact on participation and quality of life. This protocol is administered to each child at the end of the tele-rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Children with congenital or acquired brain injuries and/or neurodevelopmental disabilities
* Aged from 4-18 years old
* MACS < 5
* Cognitive functioning allowing an adequate understanding of the proposed activities and cooperation in exercises investigated by appropriate rating scales (WPPSI-III or WPPSI-IV or WISC-IV or WAIS-IV or LEITER-R or LEITER-3 or RAVEN Matrices).
* Distance from the clinical center in order to permit periodic in-person assessments
* Internet access
* Parents or legal guardians able to commit to and cooperate in an intensive home-based rehabilitation program.

Exclusion Criteria:

* Severe comorbidities and/or severe cognitive disability

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Scores of One shot feasibility questionnaire (5-point likert scale) | [Time frame: T0 (after the first assessment session with technological system (one shot))]
  An ad hoc feasibility questionnaire has been developed, according to the scientific literature, in order to investigate the acceptability and usability of the motor, cognitive, speech-communication assessment with the use of new technologies taken into account in the study. The questionnaire has been administered to the main stakeholders (clinicians, children) at the end of the one shot session assessment, delivering cognitive, motor or speech-communication activities, in order to investigate the usability and acceptability of the system with the child. Higher scores means a greater feasibility for the stakeholder who filled the questionnaire. Score ranges in the clinican form 16 to 80, while for the children form 18-90.
Tele-rehabilitation feasibility measures: Adherence to the study | [Time Frame: T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)]
  Rate of acceptance of the participation in the study calculated as the number of eligible participants that agree to join the project.
Tele-rehabilitation feasibility measures: Adherence to the training | [Time Frame: T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)]
  Total number of training sessions completed on the total number of sessions scheduled by the clinicians, expressed as a ratio.
Tele-rehabilitation feasibility measures: Number of dropouts | [Time Frame: T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)]
  Number of participants that will not complete the all study procedures.
Tele-rehabilitation feasibility measures: Number of sessions completed in the target time | [Time Frame: T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)]
  Total number of training session completed in the timeframe setted by clinicians.
Tele-rehabilitation feasibility measures: Technical problems encountered that prevent the program from running | [Time Frame: T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)]
  Number of issues and malfunctioning experimented by clinicians and families during the training sessions.
Scores of training feasibility questionnaire (5-point likert scale) | [Time Frame: T1 (at the end of the tele-rehabilitation, i.e. 3 months after the start of treatment)]
  An ad hoc feasibility questionnaire has been developed, according to the scientific literature, in order to investigate the acceptability and usability of the tele-rehabilitation training delivered through the technologies used in the study. The questionnaire has been administered to the main stakeholders (clinicians, caregivers, children) at the end of the training, in order to investigate required effort, adaptability of the training at home, exercises customization, system suidabiliy. Higher scores means a greater feasibility for the stakeholder who filled the questionnaire. Score ranges in the clinican form 20 to 100, while for the children and caregivers forms 24-120.

SECONDARY OUTCOMES:
Changes in the Sustained attention subtest of Leiter 3 | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  Sustained Attention is a subtest of the Leiter-3 non-verbal cognitive scale. It allows the assessment of visual sustained attention through barrage tasks of increasing complexity within a set time frame. The number of correctly selected target elements are recorded. Raw scores range from 0 to 217, while standardised score range from 0 to 20. Higher scores revealed better performances.
Changes in the visual attention subtest (CP) of Italian battery for ADHD (BIA) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  CP is a subtest of the Italian battery for ADHD (BIA). This subtest allows the assessment of visual sustained attention through barrage tasks of increasing complexity. Number of omissions are recorded (ranging from 0 to 54), and then converted in percentile scores. Lower raw scores reveal better performances.
Changes in the Conners' Parent Rating Scale - Brief version | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  Conner's Parent Rating Scale is a parent report questionnaire about clinical behaviours in children, with a specific focus on ADHD symptoms. Parents have to rate each item administered according to the how often this behaviour is shown by their child in the last month, circling the best option on a 3-point Likert scale. Four indices are then extracted and converted in T scores: oppositional behaviour (scores range 0 to 18), inattention/cognitive problems (scores range 0 to 18), hyperactivity (scores range 0 to 18), ADHD index (scores range 0 to 36). Higher scores reveal clinical behaviour.
Changes in the Visuo-motor precision subtest of NEPSY II | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  Visuo-motor precision is a subtest of the NEPSY II battery, used for the assessment of the ability to follow a narrow path with the pencil in an accurate and quick way. Total execution time and number of errors are recorded and then converted in percentile or standardized scores (ranging from 1 to 19). Higher scores reveal a better performance.
Changes in the Developmental Test Of Visuo-Motor Integration (VMI) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  Visuo-motor integration task is a paper and pencil test requiring geometrical figures to be copied, assessing difficulties in integrating or coordinating visual perceptual and motor (finger and hand movement) abilities. The number of figures correctly reproduced is recorded and then converted in standardized scores. Raw scores range from 0 to 27. Higher scores reveal a better performance.
Changes in the digit span forwards and backward subtests of BVN both for children aged 5-11 and for children aged 12-18 | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  Digit span is a subtest of BVN battery both for 5-11 and for 12-18 versions, allowing the assessment of short term and working memory abilities in the verbal domain though the repetition of a sequence of numbers of increasing length, following the same or a reverse order. The length of the last sequence correctly retrieved is recorded as the span, ranging from 3 to 9 in the forward condition and from 2 to 8 in the backward. Higher span reveals better performance.
Changes in the Corsi Block Tapping test subtest of BVS-Corsi | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  Corsi Block Tapping task Is a subtest of the Italian BVS-Corsi battery, assessing short term and working memory abilities in the visuo-spatial domain though the repetition of a sequence (of increasing length) of blocks tapped by examiners, following the same or a reverse order.
  The length of the last sequence correctly retrieved is recorded as the span, ranging from 3 to 8 in the forward condition and from 2 to 7 in the backward. Higher span reveals better performance.
Changes in the Behaviour Rating inventory of executive function (BRIEF 2/P ) for parents | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  Questionnaire administered to parents in order to assess executive functioning in daily life contexts. Parents have to rate each item administered according to the how often this behaviour is shown by their child in the last six months, circling the best option on a 3-point Likert scale. In the BRIEF 2 version, 9 scales are then extracted and converted in T scores: inhibition (ranging 8-24), self-monitoring (ranging 4-12), shift (ranging 8-24), emotional regulation (ranging 8-24), initiate (ranging 5-15), working memory (ranging 8-24), plan/organize (ranging 8-24), task monitoring (ranging 5-15), material organization (ranging 6-18); in the BRIEF P version, 5 scales are then extracted and converted in T scores: inhibition (ranging 16-48), shift (ranging 10-30), emotional regulation (ranging 10-30), working memory (ranging 17-51), plan/organize (ranging 10-30). Composite scores could be also calculated. Higher scores reveal clinical behaviours.
Changes in the route finding subtest of NEPSY II | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  Route finding is a subtest of the NEPSY II battery, assessing the ability to use a small schematic map to locate a target on a larger schematic map, therefore orienting in visuo-spatial coordinates. Raw scores range from 0 to 10, and then percentile scores are extracted. Higher scores reveal a better performance.
Changes in the arrow subtest of NEPSY II | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  Arrow subtest of the NEPSY II battery, assess the ability to judge lines orientation, considering and estimating direction, in distance, orientation and angularity. Raw scores range from 0 to 38, and then percentile scores are extracted. Higher scores reveal a better performance.
Changes in the Gross Motor Function Measure 88 (GMFM-88) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  The GMFM-88 assess gross motor function in children between 5 months to 16 years of age according to five dimensions: (i) Lying and Rolling, (ii) Sitting, (iii) Crawling and Kneeling, (iv) Standing, and (v) Walking, Running and Jumping. There is a four-point ordinal scoring system for each GMFM item. Then, the item scores can be summed in order to calculate raw and percentage scores for each of the five dimensions, the selected target areas, and the total GMFM-88 score. The higher the score, the better the gross motor skills.
Changes in the Assisting Hand Assessment (AHA) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  This assessment measures the assisting hand performance in children with unilateral upper limb disabilities, during bimanual performances. It can be used for children aged between 18 months and 18 years, with playful session made of semi-structured activities calibrated on the different ages (different board games). Is a standardized criterion-referenced test and the sum of scores may vary between 20 and 80, where a higher score indicates a higher ability level; the scaled score ranges between 0 and 100 and is a transformation of the sum score to a percentage distribuition within the scale, where 100 indicates that all test items were performed with the highest scores, and 0 means that all test items were performed with the lowest points.
Changes in Both Hand Assessment (BoHA) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  This assessment measures both hands performance in children with bilateral cerebral palsy, during bimanual performances. It can be used for children aged between 18 months and 12 years, with playful session made of semi-structured activities calibrated on the different ages (different board games). Is a standardized criterion-referenced test and the sum of scores may vary between 20 and 80, where a higher score indicates a higher ability level; the scaled score ranges between 0 and 100 and is a transformation of the sum score to a percentage distribuition within the scale, where 100 indicates that all test items were performed with the highest scores, and 0 means that all test items were performed with the lowest points.
Changes in the Melbourne Assessment of Unilateral Upper Limb Function o Melbourne Assessment 2 (MUUL o MA2) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  It is a valid and reliable criterion-referenced test that measures unilateral upper extremity quality of movement in children, aged 2.5 to 15 years, with neurological impairments according four elements: (i) Range of movement, (ii) Accuracy of reach and placement, (iii) Dexterity of grasp, release and manipulation and (iv) Fluency of movement. Scoring is completed across the 30 score items using a three-, four- or five-point scale and individually defined scoring criteria. Item scores relating to each element of movement measured are summed within the corresponding sub-scale. A child's final score on the MA2 is reported as four separate scores, one for each element of movement quality measured. A higher score indicates a higher upper limb ability investigated.
Changes in the Abilhand Kids | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  This questionnaire measures the manual abilities of children with CP (6-15 years old), with a particular reference to the independence in achieving some goals of everyday life, exploring if some activities are easily performed, if they present some difficulties or if they are impossible. It can be answered by parents or children and it requires 10 minutes.
Changes in the Box and Block test (BBT) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  It measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations from childhood to adults. The score is given by the number of blocks carried from one compartment to the other in one minute. Higher scores on the test indicate better gross manual dexterity. The two hands will be both tested starting from the dominant one.
Changes in the Movement Disorders - Childhood Rating Scale 4-18 revised (MD-CRS 4-18 R) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  The MD-CRS R is a standardized and validated, child-oriented rating scale aimed at describing and assessing movement disorders in children and adolescents aged 4-18 years, and their influence on activities of daily living or motor function in different regions of the body at rest and while performing specific tasks. All items are rated on a five-point ordinal scale (0-4), in which the lowest score means better performance.
Changes in the 6 minutes walk test (6MWT) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  The 6MWT assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. it can be used in preschool children (2-5 years), children (6-12 years) adults (18-64 years), elderly adults (65+) with a wide range of diagnoses including. An increase in the distance walked during 6 minute indicates improvement in basic mobility.
Changes in the Functional Reach Test (FRT) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  It is a functional assessment tool of dynamic balance evaluated in one simple task in standing position. It measures the maximum distance an individual can reach with an anterior shift with a fixed base of support. Scores are determined by assessing the difference between the start and end position is the reach distance (measured in inches or cm). Greater value (distance) = better balance and decreased falls risk. Three trials are done and average of last two noted
Changes in the Pediatric Berg Balance Scale (PBS) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  The PBS is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children with mild to moderate motor impairments. The scale consists of 14 items criterion-references that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
Changes in the Timed up and go (TUG) | [Time Frame: T0 (before beginning of the treatment); T1 (at the end of the treatment, i.e. 3 months after the start of treatment)]
  The TUG test assesses mobility, balance, walking ability, and fall risk. It is a functional dynamic balance test which measures the time it takes for the patient to stand up from a chair, walk 3 meters, turn around, walk back, and sit down.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No